CLINICAL TRIAL: NCT01628666
Title: Prevention of Arrhythmia Device Infection Trial (PADIT) Cluster Crossover Study
Brief Title: Prevention of Arrhythmia Device Infection Trial (PADIT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PADIT Cluster Crossover Study
Record Dates: First submitted 2012-06-04; First posted 2012-06-27 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Arrhythmia
Keywords: Arrhythmia; Device Procedure; Antibiotics; Infection; Cluster
MeSH Terms: conditions — Arrhythmias, Cardiac; Infections | interventions — Cefazolin; Vancomycin; Bacitracin; Cephalexin; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Experimental): Preoperative Antibiotics: Cefazolin preoperative, vancomycin in penicillin allergic patients.
  Interventions: Drug: Conventional
- Incremental (Experimental): Preoperative antibiotics (Cefazolin and Vancomycin) Bacitracin pocket wash and 2 days of oral Cefalexin post operative.
  Interventions: Drug: Incremental

INTERVENTIONS:
Drug: Incremental — Single dose of Cefazolin and Vancomycin preoperatively, bacitracin wash and cefalexin post operative.
  Other Names: Cefazolin; Vancomycin; Bacitracin; Cefalexin
  Arms: Incremental
Drug: Conventional — Cefazolin preoperative
  Other Names: Cefazolin
  Arms: Conventional

SUMMARY:
The goal of the study is to compare whether a center-wide policy of incremental antibiotic therapy will reduce CIED infection rate compared to a policy of conventional antibiotic prophylaxis in high-risk patients undergoing arrhythmia device procedures. All antibiotics used are approved for use and readily available.

DETAILED DESCRIPTION:
This is a randomized prospective cluster crossover trial to track outcomes of high infection risk patients undergoing arrhythmia device procedures. Centres will be randomized to either conventional antibiotic therapy or incremental antibiotic therapy. Patients will not be randomized. Centres will be randomized to one therapy and then cross over to the next after 6 months. At one year they will randomize again and then cross over for the final time at 18 months. During each treatment period the randomized antibiotic therapy will be used on all centre patients undergoing a device implant procedure.

Ethics approval has been obtained in all sites for waiver of consent with notification of the study (i.e. data collection is taking place to track infection rates). A third of sites obtain consent after the procedure for collection of data (but not for care, since either arm is the standard of care).

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Received one of the following procedures:

   1. A second or subsequent procedure on the arrhythmia device pocket:

      ICD, pacemaker, CRT-P, CRT-D generator and/or lead replacement
   2. Pocket or lead revision
   3. System upgrade (insertion or attempted insertion of leads)
   4. New cardiac resynchronization therapy device implant (pacemaker or ICD)
3. Patient is not known to have device infection at the time of the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12814 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Hospitalization attributed to device infection | Evaluation is one year post patient's procedure

SECONDARY OUTCOMES:
1. Proven device infection not requiring surgical intervention (medically treated device infection). | Up to one year post procedure
2. Any treatment with antibiotics for suspected device infection. | Up to one year post procedure
3. Antibiotic-related adverse events including culture or antigen proven C. difficile infection. | Up to one year post procedure
4. Prolongation of hospitalization due to proven or suspected adverse events from the antibiotic therapy. | Up to one year post procedure
Cost benefit analysis | At completion of data collection period
6. Rate of device/lead extraction 12 months post patient's procedure (regardless of the cause). | Up to one year post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krahn, MD, Principal Investigator — University of British Columbia
Locations (1):
- Coordinating Centre: Population Health Research Institute, Hamilton, Ontario, Canada